CLINICAL TRIAL: NCT05349149
Title: Role of IL-6 in Regulating Energy Stores During Recovery From an Acute Exercise Bout
Brief Title: IL-6 Regulation of Energy Stores During Recovery From an Acute Exercise Bout
Acronym: REX-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helga Ellingsgaard (Other)
Responsible Party: Sponsor-Investigator, Helga Ellingsgaard, PhD, Group leader, Centre for Physical Activity Research, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-21063697
Record Dates: First submitted 2022-04-06; First posted 2022-04-27 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Glycogen Depletion
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded to the infusion of saline or tocilizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Participants will receive one 30 min intravenous infusion of tocilizumab/Actemra® (Roche). The dose will be 8 mg/kg bodyweight or a maximum of 800mg. Tocilizumab is dissolved in 100 mL 0.9% saline.
  Interventions: Drug: Tocilizumab/Actemra® (Roche)
- Saline (Placebo Comparator): As placebo, participants will receive one 30 min intravenous infusion of 100 mL 0.9% saline.
  Interventions: Drug: Saline 9%

INTERVENTIONS:
Drug: Tocilizumab/Actemra® (Roche) — The infusion of tocilizumab will antagonize IL-6 signaling for the duration of the study, allowing us to determine the role of IL-6 in regulating energy stores following acute exercise
  Arms: Tocilizumab
Drug: Saline 9% — The infusion of saline will serve as placebo for tocilizumab, allowing us to determine the role of IL-6 in regulating energy stores following acute exercise
  Arms: Saline

SUMMARY:
The aim of the study is to investigate the role of exercise-induced IL-6 in regulating energy stores and energy metabolism during recovery after an acute exercise bout. To achieve this, 30 men will be randomized to infusion placebo or tocilizumab (IL-6 receptor antibody) combined with a 2-hour exercise bout. Stable isotope tracers will be infused to determine substrate kinetics. Indirect calorimetry will be applied to determine substrate oxidation, and muscle biopsies will be taken to determine substrate uptake and storage.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (defined as meeting the ACSM's guidelines of 2.5h per week of moderate to vigorous physical activity per week), young, healthy males will be included. Participants may be included in the study if they meet all the following criteria:

  * Age ≥ 18 years and ≤ 40 years
  * BMI < 18 and > 25 kg/m2
  * Healthy (based on screening)
  * Stable body weight for 6 months
  * ≥ 2.5h/week moderate to vigorous physical activity

Exclusion Criteria:

* • Cardiovascular disease

  * Rheumatologic disease
  * Metabolic disease
  * Elite sports or high aerobic training status (VO2max > 60 mL O2/min/kg)
  * Frequent/chronic use of medications affecting physical performance or inflammation (NSAIDS, DMARDS, corticosteroids)
  * Aspirin use >100 mg/d
  * Thyroid disease
  * Current infection
  * Aspartate amino transferase (AST) or alanine amino transferase (ALT) >2x upper normal range
  * History of carcinoma
  * History of tuberculosis
  * Ketogenic diet
  * Smoking
  * Anemia (hematocrit <33%)
  * Neutrophil count <0,5x 109/l
  * Thrombocytes <50x 109/l or bleeding disorders

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is NOT based on self-representation of gender identity
Enrollment: 30 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Change in muscle glycogen content (mmol/kg/h) | Measured at 0, 120, 180 and 360 minutes
  Comparing change in muscle glycogen in the two groups from before exercise to immediately after exercise, and after 1 hour and 4 hours of recovery
Change in muscle triglycerides content | Measured at 0, 120, 180 and 360 minutes
  Comparing change in muscle triglycerides in the two groups from before exercise to immediately after exercise, and after 1 hour and 4 hours of recovery
Change in muscle expression of glucose transporter type 4 (GLUT4) | Measured at 0, 120 and 360 min
  Comparing muscle expression of GLUT4 before and immediately after exercise and 4 hours after recovery in the two groups
Change in muscle expression of fatty acid translocase (FAT/CD36) | Measured at 0, 120 and 360 min
  Comparing muscle expression of FAT/CD36 before and immediately after exercise and 4 hours after recovery in the two groups
Change in muscle expression of muscle fatty acid binding protein (FABPm) | Measured at 0, 120 and 360 min
  Comparing muscle expression of FABPm before and immediately after exercise and 4 hours after recovery in the two groups
Change in muscle expression of fatty acid transporter 4 (FATP4) | Measured at 0, 120 and 360 min
  Comparing muscle expression of FATP4 before and immediately after exercise and 4 hours after recovery in the two groups
Change in muscle expression of glycerol transporters | Measured at 0, 120 and 360 min
  Comparing muscle expression of glycerol transporters before and immediately after exercise and 4 hours after recovery in the two groups

SECONDARY OUTCOMES:
Change in glucose rate of appearance | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing glucose rate of appearance during exercise and recovery in the two groups
Change in glucose rate of disappearance | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing glucose rate of disappearance during exercise and recovery in the two groups
Change in glucose concentration | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing glucose concentration during exercise and recovery in the two groups
Change in glucose enrichment in intramuscular glycogen | Measured at 0, 120, 180 and 360 minutes
  Comparing glucose enrichment in intramuscular glycogen during rest, exercise and recovery in the two groups
Change in intramuscular glucose concentration | Measured at 0, 120, 180 and 360 minutes
  Comparing intramuscular glucose concentration during rest, exercise and recovery in the two groups
Change in glycogen fractional synthesis rate | Measured at 0, 120, 180 and 360 minutes
  Comparing intramuscular glycogen fractional synthesis rate during rest, exercise and recovery in the two groups
Change in gylcerol rate of appearance | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing gylcerol rate of appearance during rest, exercise and recovery in the two groups
Change in gylcerol rate of disappearance | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing gylcerol rate of disappearance during rest, exercise and recovery in the two groups
Change in gylcerol concentration | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing gylcerol concentration during rest, exercise and recovery in the two groups
Change in palmitate rate of appearance | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing palmitate rate of appearance during rest, exercise and recovery in the two groups
Change in palmitate rate of disappearance | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing palmitate rate of disappearance during rest, exercise and recovery in the two groups
Change in palmitate concentration | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing palmitate kinetics during rest, exercise and recovery in the two groups
Change in palmitate oxidation | Measured at -150, -60, -45, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing palmitate oxidation during rest, exercise and recovery in the two groups
Change in intramuscular palmitate content | Measured at 0, 120, 180 and 360 minutes
  Comparing intramuscular palmitate content during rest, exercise and recovery in the two groups
Change in palmitate enrichment in intramuscular triglycerides | Measured at 0, 120, 180 and 360 minutes
  Comparing palmitate enrichment in intramuscular triglycerides during rest, exercise and recovery in the two groups
Change in intramuscular triglycerides fractional synthesis rate | Measured at 0, 120, 180 and 360 minutes
  Comparing intramuscular triglycerides fractional synthesis rate during rest, exercise and recovery in the two groups
Change in haemoglobin | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing haemoglobin during rest, exercise and recovery in the two groups
Change in haematocrit | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing haematocrit during rest, exercise and recovery in the two groups
Change in differential blood count | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing differential blood count during rest, exercise and recovery in the two groups
Change in plasma IL-6 concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma IL-6 concentration during rest, exercise and recovery in the two groups
Change in plasma TNF-alpha concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma TNF-alpha concentration during rest, exercise and recovery in the two groups
Change in plasma IL-8 concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma IL-8 concentration during rest, exercise and recovery in the two groups
Change in plasma IL-10 concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma IL-10 concentration during rest, exercise and recovery in the two groups
Change in plasma IL-1beta concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma IL-1beta concentration during rest, exercise and recovery in the two groups
Change in plasma IL-1Ra concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma IL-1Ra concentration during rest, exercise and recovery in the two groups
Change in plasma IL-4 concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma IL-4 concentration during rest, exercise and recovery in the two groups
Change in plasma sIL-6R concentration | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing plasma sIL-6R concentration during rest, exercise and recovery in the two groups
Change in insulin | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing insulin during rest, exercise and recovery in the two groups
Change in c-peptide | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing c-peptide during rest, exercise and recovery in the two groups
Change in glucagon | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing glucagon during rest, exercise and recovery in the two groups
Change in growth hormone (GH) | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing GH during rest, exercise and recovery in the two groups
Change in adrenaline | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing adrenaline during rest, exercise and recovery in the two groups
Change in noradrenaline | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing noradrenaline during rest, exercise and recovery in the two groups
Change in cortisol | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing cortisol during rest, exercise and recovery in the two groups
Change in total glucagon-like peptide-1 (GLP-1) | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing total GLP-1 during rest, exercise and recovery in the two groups
Change in active GLP-1 | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing active GLP-1 during rest, exercise and recovery in the two groups
Change in gastric inhibitory peptide (GIP) | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing GIP during rest, exercise and recovery in the two groups
Change in peptide YY (PYY) | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing PYY during rest, exercise and recovery in the two groups
Change in leptin | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing leptin during rest, exercise and recovery in the two groups
Change in triglycerides | Measured at -150, -30, 10, 30, 60, 90, 120, 130, 150, 180, 210, 240, 300 and 360 minutes
  Comparing triglycerides during rest, exercise and recovery in the two groups

OTHER OUTCOMES:
Change in muscle total antioxidant capacity (TAC) | Measured in muscle biopsies taken at 0, 120 and 360 minutes
  Comparing muscle total antioxidant capacity (TAC) at rest, after exercise and recovery in the two groups
Change in muscle superoxide levels (SOD) | Measured in muscle biopsies taken at 0, 120 and 360 minutes
  Comparing muscle superoxide levels (SOD) at rest, after exercise and recovery in the two groups
Excess post-exercise oxygen consumption | Measured at -130, 0, 60, 120, 180, 240, 300 and 360 minutes
  Comparing excess post-exercise oxygen consumption between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Centre for Physical Activity Research, Rigshospitalet Section 7641, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kistner TM, Trinh B, Mfeketo K, van Hall G, Pedersen BK, Lieberman DE, Ellingsgaard H. Myokine IL-6 activity enhances post-exercise fatty acid accumulation in skeletal muscle but does not affect glycogen resynthesis. Mol Metab. 2026 Jan;103:102283. doi: 10.1016/j.molmet.2025.102283. Epub 2025 Nov 14. PMID 41242537